CLINICAL TRIAL: NCT04834674
Title: Drug-eluting Beads Transarterial Chemoembolization Combined With Apatinib and PD-1 Antibody for the Treatment of Intrahepatic Cholangiocarcinoma That Has Progressed After Standard First-line Chemotherapy
Brief Title: DEB-TACE Combined With Apatinib and PD-1 for the Treatment of Intrahepatic Cholangiocarcinoma
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Sichuan Cancer Hospital and Research Institute (Other)
Responsible Party: Principal Investigator, Guohui Xu, Sichuan Cancer Hospital and Research Institute, Sichuan Cancer Hospital and Research Institute
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: GHX
Record Dates: First submitted 2021-04-04; First posted 2021-04-08 (Actual); Last update posted 2024-06-25 (Actual); Status verified 2024-06

CONDITIONS: Intrahepatic Cholangiocarcinoma; Transarterial Chemoembolization; Apatinib; PD-1 Antibody
MeSH Terms: conditions — Cholangiocarcinoma | interventions — apatinib

STUDY DESIGN:
Intervention Model Description: Intervention：Drug-eluting beads transarterial chemoembolization with CalliSpheres microspheres Drug: Apatinib 250mg once daily (QD) oral dosing. Drug: PD-1 antibody 200mg every 3 weeks Other Name: Programmed cell death 1 antibody
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- DEB-TACE combined with apatinib and PD-1 antibody (Experimental): The participants will receive the combined treatment of local therapy (DEB-TACE, oxaliplatin and gemcitabine), antiangiogenic therapy (apatinib), and immunotherapy (PD-1 antibody)
  Interventions: Combination Product: DEB-TACE combined with apatinib and PD-1 antibody

INTERVENTIONS:
Combination Product: DEB-TACE combined with apatinib and PD-1 antibody — combination of local therapy (DEB-TACE), antiangiogenic therapy (apatinib), and immunotherapy (PD-1 antibody)

SUMMARY:
Intrahepatic cholangiocarcinoma (ICC) is a malignant tumor of biliary epithelial cells that originates from the branches of the intrahepatic bile duct at the second level and above. Its incidence accounts for about 15%-20% of primary liver malignancies, showing a gradually increasing trend. Surgical resection is currently the main method for the treatment of ICC. However, most (60% -70%) patients are diagnosed at the advanced stage. Gemcitabine plus cisplatin is the standard first-line incurable resection recommended in international and domestic guidelines. There is not a standard second-line treatment that has progressed after standard first-line chemotherapy.

The clinical benefits of immune therapies for HCC are emerging. Early clinical data already show the safety of immune checkpoint inhibition. This study is to analyze the safety and efficacy of drug-eluting beads transarterial chemoembolization combined with apatinib and carrelizumab injection in the treatment of ICC that has progressed after standard first-line chemotherapy.

Patients who were aged 18 to 80 years with a histological or cytological diagnosis of ICC，locally advanced or multiple liver metastases, including progression after gemcitabine chemotherapy, will be enrolled in this trial.

DETAILED DESCRIPTION:
This study is a single arm, single center, open label study. It is estimated that 20 patients with intrahepatic cholangiocarcinoma which progressed after treatment with standard first-line chemotherapy in patients will be enrolled. The trial period of subjects includes screening period, treatment period and follow-up period.

The drug treatment was 200 mg of PD-1 monoclonal antibody, intravenous infusion on the first day, every 21 days as a treatment cycle; mesylate apatinib, 250 mg, oral once a day, continuous oral; DEB-TACE, the CalliSpheres + gemcitabine (800mg) and oxaliplatin were injected into the hepatic artery by routine procedure, repeated every 4-6 weeks, and administered for according to the physician in charge, DEB-TACE treatment cycles. Treatment continues until the disease progresses, intolerable toxicity occurs, new anti-tumor treatment is started, informed consent is withdrawn, follow-up is lost, death occurs or treatment termination is required。 Screening will be performed between days - 21 and - 4. Informed consent was signed up to 4 weeks prior to the first day of cycle 1 before any screening procedure or evaluation was performed and the trial was fully explained to each subject.

Baseline evaluation results must be collected prior to the first trial drug administration (day 1 of cycle 1). Baseline assessments may be performed between days - 3 and - 1 or on day 1 of cycle 1. If performed within 3 days before the first day of cycle 1, the screening results can be used as baseline results.

The tumor imaging was evaluated every 4-6 weeks since the first administration, and every 12 weeks (± 7 days) after 24 weeks. If there are clinical indications for disease progression, tumor evaluation is more frequent. In the event of disease progression, unacceptable toxicity, the subject's request to discontinue the trial or the subject's withdrawal of consent, the subject will discontinue the trial treatment.

When the trial treatment is stopped, the treatment visit shall be stopped within 7 days after the treatment is stopped in order to stop the treatment examination.

After the end of the treatment period (up to 2 years), subjects who can benefit from the study drug will continue to study the treatment of the drug until disease progression, intolerable adverse reactions, withdrawal of intensive care facility (ICF), other anti-tumor treatment, loss of follow-up, death or termination of the study.

After the occurrence of a clinical event, if it is judged by the investigators that it should be attributed to the progress of the disease and it is unlikely to recover even if the patient continues to receive treatment, it can be evaluated as clinical deterioration. It is up to the investigator to discuss and decide whether to continue or stop the treatment for the subject and record in the study file.

At the end of the study, subjects who are still under study treatment can continue to receive treatment through another extended study or other forms at the discretion of the investigator if they are stable or relieved in the efficacy evaluation and can tolerate the adverse reactions.

ELIGIBILITY:
Inclusion Criteria:

1. The diagnosis of ICC
2. Patients must have at least one tumor lesion that can be accurately measured according to mRECIST criteria.
3. Stand first-line chemotherapy resistance.
4. Performance status (PS) ≤ 2 (ECOG scale).
5. Child Pugh score ≤ 7.
6. Not amendable to surgical resection ,local ablative therapy and any other cured treatment.
7. Platelet count ≥ 50,000/μL Hemoglobin ≥ 8.5 g/dL Total bilirubin ≤ 30mmol/L Serum albumin ≥ 32 g/L ASL and AST ≤ 6 x upper limit of normal Serum creatinine ≤ 1.5 x upper limit of normal INR ≤ 1.5 or PT/APTT within normal limits Absolute neutrophil count (ANC) >1,500/mm3
8. Sign the written informed consent, and be able to follow the visit and relevant procedures specified in the plan

Exclusion Criteria:

1. Evidence of hepatic decompensation including ascites, gastrointestinal bleeding or hepatic encephalopathy
2. Known history of HIV
3. History of organ allograft
4. Known or suspected allergy to the investigational agents or any agent given in association with this trial.
5. Cardiac ventricular arrhythmias requiring anti-arrhythmic therapy
6. Evidence of bleeding diathesis.
7. Patients with clinically significant gastrointestinal bleeding within 30 days prior to study entry.
8. Known central nervous system tumors including metastatic brain disease
9. Tumor burden≥70%, diffuse liver cancer or tumor is not suitable for mRECIST standard evaluation.
10. Received local treatment (ablation therapy), surgery resection and radiotherapy for ICC before the first administration.
11. Tumor thrombus of main portal vein, or involving superior mesenteric vein at the same time.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2024-07-01 (Estimated); Primary Completion 2025-04-30 (Estimated); Study Completion 2026-04-30 (Estimated)

PRIMARY OUTCOMES:
objective response rate (ORR) | Change from baseline tumor volume at 6 months
  The proportion of patients whose tumor volume reduction reaches the predetermined value and can maintain the minimum time limit. It is the sum of the proportion of complete response (CR) and partial response(PR). That is, ORR = CR + PR
progression free survival (PFS) | Up to 24 months, from date of enrollment until the date of first documented progression or date of death from any cause, whichever came first, assessed up to 24 months
  Progression free survival period refers to the period from the beginning of treatment to the time when patients with cancer progress is observed or death occurs for any reason.

SECONDARY OUTCOMES:
overall survival (OS) | 1 year
  the time from the beginning of treatment to death caused by any reason (the last follow-up time is for the patients who lost the visit; the end of the study is for the patients who are still alive)
disease control rate (DCR) | 6 months
  It is the sum of the proportion of complete response (CR), partial response(PR) and stable disease(SD). That is, DCR = CR + PR + SD
time to progression (TTP) | Up to 24 months, from date of enrollment until the date of first documented progression or date of death from any cause, whichever came first, assessed up to 24 months
  Time from the beginning of treatment to the objective progression of tumor

CONTACTS AND LOCATIONS:
Locations (1):
- Sichuan Cancer Hospital and Research Institute, Chengdu, Sichuan, China